CLINICAL TRIAL: NCT00102700
Title: A Phase II Study of ARQ 501 in Combination With Gemcitabine in Adult Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: ARQ 501 in Combination With Gemcitabine in Subjects With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-212
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Pancreatic Cancer; Adenocarcinoma
Keywords: cancer; solid tumor; advanced solid tumor; pancreas; pancreatic cancer; cancer of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasms | interventions — beta-lapachone; Gemcitabine

INTERVENTIONS:
Drug: ARQ 501 in combination with gemcitabine

SUMMARY:
The study will document the safety and efficacy of the combination of ARQ 501 and gemcitabine in patients with treatment-naïve, unresectable, metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized study of ARQ 501 in combination with gemcitabine in adult patients with treatment-naïve, unresectable, metastatic pancreatic adenocarcinoma. The study objectives are:

Primary Objective:

* Assess the overall response rate (ORR) of patients treated with ARQ 501 in combination with gemcitabine.

Secondary Objectives:

* Determine time to tumor progression (TTP) of patients treated with ARQ 501 in combination with gemcitabine
* Further characterize the safety of ARQ 501 in combination with gemcitabine

ELIGIBILITY:
Inclusion Criteria:

* Have a pathologically confirmed diagnosis of unresectable, metastatic pancreatic adenocarcinoma
* Be treatment-naïve.
* Have measurable disease per RECIST Criteria.
* Be ≥18 years old.
* Have a Karnofsky Performance Status (KPS) of ≥70%.
* Have an estimated life expectancy of ≥12 weeks.
* Be male or a non-pregnant, non-lactating female patient. Patients who are fertile agree to use an effective barrier method of birth control (e.g., latex condom, diaphragm, or cervical cap) to avoid pregnancy.
* Have a negative serum or urine pregnancy test within 7 days prior to the first dose of study drug (if patient is a female of childbearing potential).
* Sign a written informed consent form.
* Have adequate organ function as indicated by acceptable laboratory values obtained within 7 days prior to the first dose of study drug.

Exclusion Criteria:

* Have received any prior therapy for the treatment of their pancreatic malignancy (including chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational).
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
* Are pregnant or lactating.
* Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
* Have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Have symptomatic or untreated central nervous system (CNS) metastases.
* Have a known hypersensitivity to gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Document progression free survival after treatment with ARQ 501 and gemcitabine

SECONDARY OUTCOMES:
Document safety and efficacy of ARQ 501 in combination with gemcitabine

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of South Alabama, Mobile, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Scripps Cancer Center, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Unversity of Kentucky Medical Center - Markey Center, Lexington, Kentucky
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jeffrey Meyerhardt, Boston, Massachusetts
  - Jacobi Medical Center, The Bronx, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Virginia Cancer Institute, Richmond, Virginia